CLINICAL TRIAL: NCT05163392
Title: A Silver Lining in the VAD Sky: Impact of Silver Dressing on LVAD Associated Driveline Infection
Brief Title: A Silver Lining in the VAD Sky
Acronym: LVAD-SilverD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: International Consortium of Circulatory Assist Clinicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-35805
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: LVAD (Left Ventricular Assist Device) Driveline Infection

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of 2 arms conducted in parallel.
  The trial arm kits include:
  1. For standard dressing: a silverlon antimicrobial patch, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be weekly.
  2. For sensitive skin dressing: a silverlon antimicrobial patch, Providone/iodine swabs for cleaning, an occlusive dressing with window, and sensitive driveline anchors. The driveline dressing change frequency will be weekly.
  The control arm kits include:
  1. For standard dressing: No antimicrobial barrier, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96 hours.
  2. For sensitive skin dressing: No antimicrobial barrier, Providone/iodine swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96hr.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SilverD (Experimental): The SIlverD arm includes:
  1. For standard dressing: a silverlon antimicrobial patch, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be weekly.
  2. For sensitive skin dressing: a silverlon antimicrobial patch, Providone/iodine swabs for cleaning, an occlusive dressing with window, and sensitive driveline anchors. The driveline dressing change frequency will be weekly.
  Interventions: Device: Silverlon
- ControlD (Active Comparator): The ControlD arm includes:
  1. For standard dressing: No antimicrobial barrier, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96 hours.
  2. For sensitive skin dressing: No antimicrobial barrier, Providone/iodine swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96hr.
  Interventions: Device: Control

INTERVENTIONS:
Device: Silverlon — SIlver-plated biopatch
  Arms: SilverD
Device: Control — Tegaderm without biopatch
  Arms: ControlD

SUMMARY:
The investigators propose to conduct a prospective randomized trail (RCT) of a driveline management protocol. The study will be initiated at UCSF from January 1st 2022 to December 31st 2022 as a pilot to be extended to other sites with the ultimate goal to develop a multi-center RCT. The driveline dressing protocol studied will include a silver-based dressing barrier as well as a dressing change protocol and material designed to reduce the risk of driveline dressing induced dermatitis and allergies. Assessment will include DLI rates, DLI speciation, dermatitis rate, comfort, ease of use, compliance and cost

DETAILED DESCRIPTION:
This prospective research clinical trial will be conducted in a single academic medical center. The enrollment period will be between January 1st, 2022 and December 31st, 2023. The initial follow-up period will be closed on December 31st 2023 with a continuation of the follow-up until December 31st 2024. Patients will be selected from current LVAD patients followed by our medical center clinic and from patients implanted with LVAD at our center during the study enrollment timeframe. Patients will be randomly assigned to the control protocol and the silver protocol. Both protocols will be taught to the patients and nursing staff by the VAD coordinators. The comparative evaluation will be done through adverse event collection, driveline culture results, patient survey and DL photos at specific intervals.

Interventions A new driveline dressing kit will be trialed on patients randomized to the intervention arm of the study. Both arms will have a regular dressing kit and a sensitive dressing kit.

The trial arm kits include:

1. For standard dressing: a silverlon antimicrobial patch, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be weekly.
2. For sensitive skin dressing: a silverlon antimicrobial patch, Providone/iodine swabs for cleaning, an occlusive dressing with window, and sensitive driveline anchors. The driveline dressing change frequency will be weekly.

The control arm kits include:

1. For standard dressing: No antimicrobial barrier, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96 hours.
2. For sensitive skin dressing: No antimicrobial barrier, Providone/iodine swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96hr.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Implanted with LVAD as DT or BTT at the Academic Medical Center with implantation scheduled between January 1st, 2022 and December 31st, 2022

Exclusion Criteria:

* A history of DLI
* A history of sternal wound infection
* Implantation secondary to VAD exchange for device infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Klein, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Only aggregate data might be shared.

REFERENCES:
- [Background] Kusne S, Mooney M, Danziger-Isakov L, Kaan A, Lund LH, Lyster H, Wieselthaler G, Aslam S, Cagliostro B, Chen J, Combs P, Cochrane A, Conway J, Cowger J, Frigerio M, Gellatly R, Grossi P, Gustafsson F, Hannan M, Lorts A, Martin S, Pinney S, Silveira FP, Schubert S, Schueler S, Strueber M, Uriel N, Wrightson N, Zabner R, Huprikar S. An ISHLT consensus document for prevention and management strategies for mechanical circulatory support infection. J Heart Lung Transplant. 2017 Oct;36(10):1137-1153. doi: 10.1016/j.healun.2017.06.007. Epub 2017 Jun 23. No abstract available. PMID 28781010
- [Background] Koken ZO, Yalcin YC, van Netten D, de Bakker CC, van der Graaf M, Kervan U, Verkaik NJ, Caliskan K. Driveline exit-site care protocols in patients with left ventricular assist devices: a systematic review. Eur J Cardiothorac Surg. 2021 Sep 11;60(3):506-515. doi: 10.1093/ejcts/ezab195. PMID 33963835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 patients were enrolled and all met inclusion criteria and were randomized to treatment or placebo
Groups:
- SilverD: The SIlverD arm includes:
  1. For standard dressing: a silverlon antimicrobial patch, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be weekly.
  2. For sensitive skin dressing: a silverlon antimicrobial patch, Providone/iodine swabs for cleaning, an occlusive dressing with window, and sensitive driveline anchors. The driveline dressing change frequency will be weekly.
  Silverlon: SIlver-plated biopatch
- ControlD: The ControlD arm includes:
  1. For standard dressing: No antimicrobial barrier, CHG swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96 hours.
  2. For sensitive skin dressing: No antimicrobial barrier, Providone/iodine swabs for cleaning, an occlusive dressing with window, and driveline anchors. The driveline dressing change frequency will be every 96hr.
  Control: Tegaderm without biopatch
Period: Overall Study
Arm/Group | SilverD | ControlD
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SilverD | ControlD | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15) | 45 (14) | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 14 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 25
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.8 (4.6) | 38.4 (5.1) | 34.28 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Driveline Infection Rate
Description: Number of driveline infection per 100 patient-months
Time Frame: 2 year
Measure: Number; unit: infections per 100 patient-month
Arm/Group | SilverD | ControlD
Number analyzed (Participants) | 14 | 11
infections per 100 patient-month | 0.51 | 06.28

2. Secondary Outcome: Time to First Driveline Infection
Description: Number of days to first driveline infection
Time Frame: 2 year
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | SilverD | ControlD
Number analyzed (Participants) | 14 | 11
days | 458 [279 to 637] | 232 [74 to 390]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 1 year
Description: 5 patients died due to heart failure. Cause of death was unrelated to the study.
Arm/Group | SilverD | ControlD
All-Cause Mortality (participants affected / at risk) | 3/14 | 2/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05163392/Prot_SAP_ICF_003.pdf